CLINICAL TRIAL: NCT04705259
Title: A Multimodal Intervention to Optimise Antimicrobial Use in Residential Aged Care Facilities (ENGAGEMENT Study): Protocol for a Stepped Wedge Cluster Randomised Trial
Brief Title: A Multimodal Intervention to Optimise Antimicrobial Use in Residential Aged Care Facilities (ENGAGEMENT Study)
Acronym: ENGAGEMENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Queensland (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020002193
Record Dates: First submitted 2020-12-03; First posted 2021-01-12 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2020-11

CONDITIONS: Antimicrobial Stewardship; Antibiotics Causing Adverse Effects in Therapeutic Use
Keywords: Antimicrobial stewardship; Antibiotic prescribing; Aged care

STUDY DESIGN:
Intervention Model Description: Stepped wedge randomised control study
Masking Description: Education intervention where the facilities will be made aware of best practice guidelines and protocols with respect to antibiotic prescribing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENGAGEMENT bundle (Active Comparator): A multimodal bundle of interventions to optimise antibiotic prescribing in residential aged care facilities. The bundle includes education for nurses and general practitioners caring for residents, telehealth support and implementation of state-wide guidelines.
  Interventions: Behavioral: Antimicrobial Stewardship ENGAGEMENT bundle
- Usual care (Placebo Comparator): Usual facility practices with regards to antibiotic prescribing and review
  Interventions: Behavioral: Antimicrobial Stewardship ENGAGEMENT bundle

INTERVENTIONS:
Behavioral: Antimicrobial Stewardship ENGAGEMENT bundle — Given that a single intervention is unlikely to be effective in stewardship programs, nor in care improvement processes at RACFs [7], this trial will deliver a set of multimodal, multidisciplinary interventions to optimise antibiotic use in RACFs. This RACF AMS ENGAGEMENT bundle will comprise the following key interventions:
  * Education and engagement of prescribers, nurses, pharmacists and residents and family members
  * Nursing initiatives to improve UTI diagnosis and reduce inappropriate urine testing
  * Guideline development specific to antibiotic use in RACF residents
  * Antimicrobial stewardship team creation in RACF with GP involvement
  * EMergency department liaison and use of clinical pathways to ensure consistency of practice across the care continuum
  * ElectroNic decision support to guide RACF urine testing and GP antibiotic prescribing
  * Telehealth support for key intervention components

SUMMARY:
The antimicrobial stewardship ENGAGEMENT study aims to deliver a bundle of interventions, including education of GPs and nursing staff, guideline implementation and telehealth support for 18 residential aged care facilities (RACFs) in Queensland Australia to help optimise antibiotic prescribing and reduce inappropriate use. The trial will involve 18 licenced RACFs with 50 or more residents and is set to commence in June 2021.

DETAILED DESCRIPTION:
INTRODUCTION Inappropriate antibiotic use can cause harm and promote antimicrobial resistance, which has been declared a major health challenge by the World Health Organisation. In Australian Residential Aged Care Facilities (RACFs), the most common indications for antibiotic prescribing are for suspected infections of the urinary tract, respiratory tract, and skin and soft tissue. Studies indicate that a high proportion of these prescriptions are noncompliant with best prescribing guidelines. To date a variety of interventions have been reported to address inappropriate prescribing and overuse of antibiotics but with mixed outcomes. The present study aims to identify the impact of a set of sustainable, multi-modal interventions in residential aged care targeting three common infection types, using a robust methodology.

METHODS AND ANALYSIS This study will be conducted using a stepped-wedge cluster randomised trial that will recruit 18 RACFs (each RACF will be considered as one cluster), over a 20 month observation period. Initially an antimicrobial stewardship needs assessment toolkit will be piloted in seven RACFs from different service providers. This will enable the refinement and targeted implementation of the intervention bundle, based on existing requirement of facilities. A multimodal multi-disciplinary set of interventions, the 'ENGAGEMENT bundle', will be tailored to the needs of facilities. This bundle will be implemented as part of the stepped wedge randomised control trial. The key elements of the intervention bundle include education for nurses and general practitioners, telehealth support and formation of an antimicrobial stewardship team. Prior to the sequential introduction of the intervention, each site will act as its own control, in relation to usual care processes for antibiotic use and stewardship.

The primary outcome for this study will be antibiotic consumption measured using defined daily doses (DDDs). Cluster-level rates will be calculated using total occupied bed numbers within each RACF during the post-randomisation observation period as the denominator. Results will be expressed as rates per 1000 occupied bed days. An economic analysis will be conducted to compare the costs associated with the intervention to that of usual care.

ELIGIBILITY:
Eligibility is at the Residential Aged Care Facility (RACF) level. If the facility is eligible to participate de-identified data from all facility residents will be included for the duration of the the study.

Inclusion Criteria:

* All residents of RACFs with at least 50 residents
* RACFs located in South East Queensland, Australia

Exclusion Criteria:

* RACFs with less than 50 residents;
* RACFs unable to provide reports for baseline data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-12-24 (Estimated)

PRIMARY OUTCOMES:
Defined Daily Doses (DDDs) of Antibiotics | 18 months
  The primary outcome measure for this trial is antibiotic use as measured by DDDs of antibiotics per 1000 resident bed days.

SECONDARY OUTCOMES:
Urine Samples | 18 months
  Number of urine samples collected per 1000 resident bed days between the control vs intervention periods
Susceptibility of pathogens | 18 months
  Percent susceptibility of Enterobacteriaceae to ceftriaxone, ciprofloxacin, cephalexin and amoxicillin-clavulanate measured using antibiograms
All cause on-year mortality | 18 months
  All-cause on-year mortality rates of residential aged care facility (RACF) residents between the control vs intervention periods (per 1000 resident bed days and median rate across facilities)
Hospital admissions | 18 months
  Number of RACF residents admitted to hospital during the control vs intervention periods (per 1000 resident bed days and median rate across facilities)

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Bethany Christian Care, Eight Mile Plains, Queensland
  - Carinity Aged Care, Mitchelton, Queensland
  - Beaumont Care, Rothwell, Queensland
  - Vacenti Aged Care, Upper Mount Gravatt, Queensland

REFERENCES:
- [Derived] Falconer N, Paterson DL, Peel N, Welch A, Freeman C, Burkett E, Hubbard R, Comans T, Hanjani LS, Pascoe E, Hawley C, Gray L. A multimodal intervention to optimise antimicrobial use in residential aged care facilities (ENGAGEMENT): protocol for a stepped-wedge cluster randomised trial. Trials. 2022 May 21;23(1):427. doi: 10.1186/s13063-022-06323-8. PMID 35597993